CLINICAL TRIAL: NCT04300309
Title: Multicenter, Open-label, Single-arm Study to Evaluate the PK, Safety, Tolerability and Efficacy of a New Artemether:Lumefantrine (2.5 mg:30 mg) Dispersible Tablet in the Treatment of Infants and Neonates <5 kg Body Weight With Acute Uncomplicated Plasmodium Falciparum Malaria
Brief Title: Pharmacokinetics, Safety, Tolerability and Efficacy of a New Artemether-lumefantrine Dispersible Tablet in Infants and Neonates <5 kg Body Weight With Acute Uncomplicated Plasmodium Falciparum Malaria
Acronym: CALINA
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Medicines for Malaria Venture (Other); Groupe de Recherche Action en Sante (Other); Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCOA566B2307; PACTR202004535453508 (Other: PACTR)
Record Dates: First submitted 2020-02-18; First posted 2020-03-09 (Actual); Results first posted 2024-10-03 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Plasmodium falciparum; malaria; artemether; lumefantrine; neonates; infants
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- artemether lumefantrine (2.5 mg:30 mg) (Experimental): Artemether-lumefantrine (5 mg:60 mg) twice daily for 3 days
  Interventions: Drug: artemether:lumefantrine (2.5 mg:30 mg)

INTERVENTIONS:
Drug: artemether:lumefantrine (2.5 mg:30 mg) — Two oral dispersible tablets twice daily for three consecutive days. Each tablet contained artemether-lumefantrine 2.5 mg:30 mg.

SUMMARY:
The purpose of this study was to evaluate PK, safety, tolerability and efficacy of a new formulation of artemether-lumefantrine dispersible tablet in neonates and infants <5 kg body weight with acute uncomplicated Plasmodium falciparum malaria.

DETAILED DESCRIPTION:
This was a multicenter, open-label, single-arm, adaptive design with dose adaptation (deescalation or escalation) study in infants and neonates <5 kg body weight with P. falciparum malaria. There were two sequential and age-descending cohorts of participants, all <5 kg: Cohort 1 of infants >28 days of age, and Cohort 2 of neonates ≤ 28 days of age.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female neonates/infants
2. Body weight <5 kg but ≥ 2 kg
3. In Cohort 1, infants aged >28 days; in Cohort 2, neonates aged 1 to ≤28 days (3 subgroups: 1-7 days; 8-14 days; 15-28 days)
4. Microscopically confirmed diagnosis of P. falciparum malaria (or mixed infections):

   * in Cohort 1 of ≥500 and <100,000 parasites/µL asexual P. falciparum parasitemia
   * in Cohort 2 of ≥100 and <100,000 parasites/µL asexual P. falciparum parasitemia
   * either congenital or neonatal
   * either symptomatic or asymptomatic

Exclusion Criteria:

1. Head circumference < - 2 SD z-score in cm following WHO age and sex-specific reference curves (suspicion of microcephaly)
2. Presence of severe malaria (according to WHO 2015 definition)
3. HIV status :

   * in Cohort 1, patient's or patient's mother's current treatment with ARV
   * in Cohort 2, mother's known HIV positive status at patient's birth or mother's current treatment with ARV
4. Presence of the following signs of a critical condition: apnea-bradycardia, sustained bradycardia, tachycardia, desaturation, hypotension, hypothermia; or other severely deteriorated general condition (based on IMCI criteria in sick infants) (WHO 2005)
5. Presence of any clinically significant neurological condition:

   * any episode of convulsion during the present illness (in keeping with the IMCI list of general danger signs)
   * known neurological disorders (e.g. chronic seizure disorders, cerebral palsy)
6. Presence of clinically significant abnormality of the hepatic and renal systems
7. Patients unable to swallow or whose drinking is impaired
8. Known hypersensitivity of the patient or either patient's parent to artemether, lumefantrine, any of the excipients of Coartem®/Riamet® Dispersible tablet, or to drugs of similar chemical classes
9. History of malabsorption or previous gastrointestinal surgery, or history of radiation therapy that could affect drug absorption or metabolism, or any other disorder or history of a condition that could interfere with drug absorption, distribution, metabolism, or excretion
10. Known family history of congenital prolongation of the QTc interval or sudden death or with any other clinical condition known to be associated with prolongation of the QTc interval such as history of symptomatic cardiac arrhythmias, with clinically relevant bradycardia or with severe cardiac disease
11. Disturbances of electrolyte balance (e.g. hypokalaemia or hypomagnesaemia)
12. Presence of any age-adjusted clinically or hematologically relevant laboratory and blood chemistry abnormalities
13. Patients who received any antimalarial drug, including antibiotics with antimalarial activity, within 14 days of trial start, or any other prohibited drug (see Table 6-2)
14. Patients who received an investigational drug within 5 half-lives of enrollment or participated in an investigational study or within 30 days, whichever is longer

Max Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-07-02 (Actual); Study Completion 2024-05-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Burkina Faso (2):
  - Novartis Investigative Site, Nanoro
  - Novartis Investigative Site, Ouagadougou
- Novartis Investigative Site, Kisantu, Bas Kongo, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wounounou G, Tiono AB, Ogutu B, Manyando C, Sagara I, Schneitter S, Bassat Q, Gaaloul ME, Marrast AC, Demin I, Winnips C, Risterucci C, Hugot S, Hofstetter G, Qian Z, Su G, Zhang J, Renner KC, Cousin M, Venishetty VK, Sayyed S, Gandhi P, Kabore B; CALINA study group. Pharmacokinetics, safety and efficacy of an optimized dose of artemether-lumefantrine in the treatment of acute uncomplicated Plasmodium falciparum malaria in neonates and infants of less than 5 kg body weight: a multicentre, open-label, single-arm phase 2/3 study (CALINA). Trop Med Health. 2025 Nov 6;53(1):151. doi: 10.1186/s41182-025-00828-z. PMID 41199347
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2407
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=676

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 3 investigative sites in 2 countries.
Pre-assignment Details: The Screening procedures began once the study informed consent had been obtained. Screening was performed within 12 hours before the first study drug administration.
Groups:
- Cohort 1: Infants >28 days of age treated with artemether-lumefantrine (5 mg:60 mg) twice daily for 3 days
- Cohort 2: Term neonates 1-28 days of age treated with artemether-lumefantrine (5 mg:60 mg) twice daily for 3 days
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started (All patients enrolled in the study) | 22 | 6
Full Analysis Set (FAS) (All patients that received any study treatment and had P. falciparum present at Screening visit) | 22 | 6
Per-Protocol Set (PPS) (Patients in the FAS who met the following criteria: a) Did not have important protocol deviations affecting efficacy; b) Took at least 80% of study medication; c) PCR corrected cure status at Day 29 could be defined.) | 17 | 6
PK Set (Patients in the FAS who had evaluable pharmacokinetics (PK) parameter data) | 22 | 6
Completed treatment phase | 22 | 6
Completed Core follow-up (43 days) | 22 | 6
Completed (Completed long-term follow up) | 21 | 6
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 22 | 6 | 28
Age, Continuous [Median (Full Range); unit: days] | 96.0 [53.0 to 157.0] | 22.5 [1.0 to 26.0] | 83.0 [1.0 to 157.0]
Age, Customized [Count of Participants; unit: Participants]
  1-7 days | 0 | 1 | 1
  8-14 days | 0 | 0 | 0
  15-28 days | 0 | 5 | 5
  >28 days | 22 | 0 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 18
  Male | 7 | 3 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 22 | 6 | 28
Weight [Median (Full Range); unit: kilograms] | 4.82 [3.89 to 4.98] | 3.50 [2.80 to 4.24] | 4.76 [2.80 to 4.98]
Plasmodium species [Count of Participants; unit: Participants] — Parasitemia determinations were performed in peripheral blood. Microscopic species determination was confirmed with polymerase chain reaction (PCR)-based methods. The assessments were performed at a central reference laboratory.
  Participants
    P. falciparum asexual forms | 21 | 6 | 27
    P. falciparum gametocytes | 4 | 1 | 5
    P. vivax | 0 | 0 | 0
    P. ovale | 0 | 0 | 0
    P. malariae | 1 | 0 | 1
    P. knowlesi | 0 | 0 | 0
Plasmodium falciparum density [Median (Full Range); unit: parasites/µL] — Parasitemia determinations were performed in peripheral blood. Giemsa stained thick fields were examined at a central reference laboratory. The parasite density was calculated according to the following formula: (number of Plasmodium falciparum parasites * actual leukocytes)/number of leucocytes counted (200 thick films fields examined)
  parasites/µL | 8400 [748 to 156400] | 3660 [384 to 52700] | 7020 [384 to 156400]

OUTCOME MEASURES:

1. Primary Outcome: Artemether Cmax After First Dose
Description: Artemether Cmax represents the highest concentration between the concentrations at 1 hour and 2 hours after first dose.
  Pharmacokinetic (PK) parameters were calculated by non-compartmental analysis based on artemether plasma concentrations.
Time Frame: 1 and 2 hours after first dose (Day 1)
Population: Participants in the PK set who had an available value for the outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 20 | 5
ng/mL | 68.0 [45.1 to 103] | 62.2 [33.6 to 115]

2. Secondary Outcome: Lumefantrine Day 8 Concentration (C168h)
Description: Pharmacokinetic (PK) parameters were calculated by non-compartmental analysis based on lumefantrine plasma concentrations.
  Dosing times were 0, 8, 24, 36, 48 and 60 hours.
Time Frame: 168 hours after first dose (corresponding to 108 hours after last dose)
Population: Participants in the PK set who had an available value for the outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
ng/mL | 353 [250 to 498] | 480 [265 to 870]

3. Secondary Outcome: Lumefantrine Cmax After Last Dose
Description: Lumefantrine Cmax represents the highest concentration among four sampling time points after last dose.
  Pharmacokinetic (PK) parameters were calculated by non-compartmental analysis based on lumefantrine plasma concentrations.
  Dosing times were 0, 8, 24, 36, 48 and 60 hours.
Time Frame: 62, 66, 68 and 84 hours after first dose (corresponding to 2, 6, 8 and 24 hours after last dose)
Population: Participants in the PK set who had an available value for the outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
ng/mL | 3180 [2530 to 4000] | 3510 [1880 to 6540]

4. Secondary Outcome: DHA Cmax After First Dose
Description: Dihydroartemisinin (DHA) is an active metabolite of artemether. DHA Cmax represents the highest concentration between the concentrations at 1 hour and 2 hours after first dose.
  Pharmacokinetic (PK) parameters were calculated by non-compartmental analysis based on DHA plasma concentrations.
Time Frame: 1 and 2 hours after first dose (Day 1)
Population: Participants in the PK set who had an available value for the outcome measure.
Measure: Geometric Mean (90% Confidence Interval); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 20 | 5
ng/mL | 11.5 [7.58 to 17.4] | 15.7 [8.53 to 28.9]

5. Secondary Outcome: Parasite Clearance Time (PCT)
Description: PCT is defined as time from the first dose until the first total and continued disappearance of asexual parasite forms which remained at least a further 48 hours. PCT is based on uncorrected parasite counts.
  Patients who received rescue medication before parasite clearance were censored at the first use of rescue medication.
  Patients without parasite clearance were censored at the time of last parasite assessment.
  PCT was calculated using the Kaplan-Meier method.
Time Frame: Up to 48 hours after first dose
Population: Full Analysis Set (FAS)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
hours | 35.0 [24.0 to 35.8] | 30.6 [23.8 to 47.6]

6. Secondary Outcome: Fever Clearance Times (FCT)
Description: FCT is defined as time from the first dose until the first time the axillary body temperature decreased below and remained below 37.5°C axillary or 38.0°C oral/tympanic/rectal for at least a further 24 hours.
  Patients who received rescue medication before fever clearance were censored at the first use of rescue medication.
  Patients without fever clearance were censored at the time of last parasite assessment.
  FCT was calculated using the Kaplan-Meier method.
Time Frame: Up to 36 hours after first dose
Population: Participants in the Full Analysis Set (FAS) who had fever at baseline
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 4 | 1
hours | 15.7 [3.9 to 29.7] | 7.6 [7.6 to 7.6]

7. Secondary Outcome: PCR-corrected Adequate Clinical and Parasitological Response (ACPR) - PPS Analysis
Description: PCR-corrected ACPR, defined as the absence of parasitemia, was evaluated on Days 15, 29 and 43. Microscopic species identification was confirmed and determined by polymerase chain reaction (PCR) genotyping methods to establish malaria recrudescence/reinfection.
  A participant was considered as PCR-corrected ACPR if the participant did not meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure and had absence of parasitemia on Days 15, 29 or 43 irrespective of axillary temperature unless the presence of parasitemia after 7 days was due to reinfection based on PCR. A presence of parasitemia after 7 days of treatment initiation was considered as a reinfection only if the parasitemia was clear before Day 8 and none of the parasite strain(s) detected on Day 8 or later matched with the parasite strain at baseline based on PCR.
Time Frame: Days 15, 29 and 43
Population: Per-Protocol Set (PPS). Five patients in Cohort 1 were excluded from the PPS due to the use of prohibited concomitant medication, i.e. erythromycin.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 17 | 6
percentage of participants
  Day 15 | 100 [80.49 to 100] | 100 [54.07 to 100]
  Day 29 | 100 [80.49 to 100] | 100 [54.07 to 100]
  Day 43 | 94.1 [71.31 to 99.85] | 100 [54.07 to 100]

8. Secondary Outcome: PCR-corrected Adequate Clinical and Parasitological Response (ACPR) - FAS Analysis
Description: as for outcome 7
Time Frame: Days 15, 29 and 43
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
percentage of participants
  Day 15 | 100 [84.56 to 100] | 100 [54.07 to 100]
  Day 29 | 95.5 [77.16 to 99.88] | 100 [54.07 to 100]
  Day 43 | 90.9 [70.84 to 98.88] | 100 [54.07 to 100]

9. Secondary Outcome: PCR-uncorrected Adequate Clinical and Parasitological Response (ACPR)
Description: PCR-uncorrected ACPR, defined as the absence of parasitemia, was evaluated on Days 8, 15, 29 and 43.
  A participant was considered as PCR-uncorrected ACPR if the participant did not meet any of the criteria of early treatment failure, late clinical failure or late parasitological failure and had absence of parasitemia on Days 8, 15, 29 or 43 irrespective of axillary temperature.
Time Frame: Days 8, 15, 29 and 43
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
percentage of participants
  Day 8 | 100 [84.56 to 100] | 100 [54.07 to 100]
  Day 15 | 100 [84.56 to 100] | 100 [54.07 to 100]
  Day 29 | 77.3 [54.63 to 92.18] | 100 [54.07 to 100]
  Day 43 | 63.6 [40.66 to 82.80] | 100 [54.07 to 100]

10. Secondary Outcome: Number of Participants With Recrudescence Events
Description: Recrudescence is defined as appearance of asexual parasites after clearance of initial infection with a genotype identical to that of parasites present at baseline. Recrudescence had to be confirmed by PCR analysis.
Time Frame: Days 15, 29 and 43
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
Participants
  Day 15 | 0 | 0
  Day 29 | 1 | 0
  Day 43 | 1 | 0

11. Secondary Outcome: Number of Participants With New Infections Events
Description: New infection is defined as appearance of asexual parasites after clearance of initial infection with a genotype different from those parasites present at baseline. New infection had to be confirmed by PCR analysis.
Time Frame: Days 15, 29 and 43
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
Participants
  Day 15 | 0 | 0
  Day 29 | 4 | 0
  Day 43 | 2 | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Number of participants with adverse events (any AEs regardless of seriousness), including changes in laboratory results qualifying and reported as adverse events.
Time Frame: From first dose of study treatment until Day 43
Population: Safety Set, including all patients who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
Participants | 17 | 4

13. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with serious adverse events (SAEs), including changes in laboratory results qualifying and reported as serious adverse events.
Time Frame: From first dose of study treatment until 12 months of age (assessed up to maximum 1 year)
Population: Safety Set, including all patients who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 22 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected from first dose of study treatment until Day 43. Deaths and serious adverse events were collected from first dose of study treatment until 1 year of age (assessed up to maximum 1 year).
Description: Adverse events are assessed in the Safety Set, including all patients who received at least one dose of study treatment.
Groups:
- Pooled Cohort: All infants and neonates who received at least one dose of artemether-lumefantrine
Arm/Group | Cohort 1 | Cohort 2 | Pooled Cohort
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/6 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/6 | 0/28
Other Adverse Events (participants affected / at risk) | 17/22 | 4/6 | 21/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=22) | Cohort 2 (N=6) | Pooled Cohort (N=28)
Anaemia (Blood and lymphatic system disorders) | 7 | 1 | 8
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 6 | 1 | 7
Pyrexia (General disorders and administration site conditions) | 8 | 2 | 10
Bacterial rhinitis (Infections and infestations) | 2 | 0 | 2
Ear infection (Infections and infestations) | 0 | 1 | 1
Gastrointestinal fungal infection (Infections and infestations) | 0 | 1 | 1
Malaria (Infections and infestations) | 9 | 0 | 9
Rhinitis (Infections and infestations) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT04300309/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04300309/SAP_001.pdf